CLINICAL TRIAL: NCT06297486
Title: A Phase 3, Single-arm, Open-label, Multicenter Study of the Safety and Efficacy of Dirloctocogene Samoparvovec (SPK 8011, Adeno-associated Viral Vector With B-domain Deleted Human Factor VIII Gene) in Adults With Severe or Moderately Severe Hemophilia A
Brief Title: Study of a Gene Therapy Treatment for Hemophilia A
Acronym: KEYSTONE 1
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Strategic Decision
Sponsor: Spark Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPK-8011-302; 2023-504537-46 (EudraCT Number)
Record Dates: First submitted 2024-02-29; First posted 2024-03-07 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Hemophilia A
Keywords: Dirloctocogene samoparvovec; SPK 8011; Blood coagulation factor VIII; FVIII; AAV-Spark200-BDD-hFVIII; Gene Therapy
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Intervention Model Description: Participants will be assigned into one of three cohorts, each receiving the same study treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A (Primary Cohort) (Experimental): Participants with severe or moderately severe hemophilia A without FVIII inhibitors using routine FVIII prophylaxis
  Interventions: Genetic: SPK-8011
- Cohort B (Experimental): Participants with severe or moderately severe hemophilia A without FVIII inhibitors using on-demand FVIII replacement therapy
  Interventions: Genetic: SPK-8011
- Cohort C (Experimental): Participants with severe or moderately severe hemophilia A without FVIII inhibitors using emicizumab prophylaxis
  Interventions: Genetic: SPK-8011

INTERVENTIONS:
Genetic: SPK-8011 — Participants will receive a single dose of SPK-8011, administered by intravenous (IV) infusion, on Day 1.
  Other Names: AAV-Spark200-BDD-hFVIII; Dirloctocogene samoparvovec

SUMMARY:
The purpose of this study is to evaluate the efficacy of SPK-8011 in preventing bleed episodes compared with FVIII prophylaxis in participants with hemophilia A without FVIII inhibitors on routine FVIII prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* Have a negative anti-AAV-Spark200 neutralizing antibody (NAb) test result.
* Are adult males with severe or moderately severe hemophilia A, defined as endogenous FVIII activity ≤3%, as documented by a certified laboratory (historically or during the Screening Period) and where the FVIII:C level is measured more than 96 hours after the prior dose of an extended-half-life FVIII
* Have ≥150 documented exposure days to an FVIII protein product such as recombinant, plasma-derived, or extended half-life FVIII product
* Have no prior history of hypersensitivity or anaphylaxis associated with the administration of any FVIII product.
* Have screening hepatic ultrasound without evidence of cirrhosis and no laboratory or clinical evidence per the Investigator's judgment of advanced liver disease or cirrhosis.
* Have a negative test for inhibitor against FVIII (ie, <0.6 Bethesda units [BU]) during screening.
* Have no documented FVIII inhibitor (ie, <0.6 BU), FVIII half-life <6 hours, or FVIII recovery <66% in the 5 years prior to screening.
* Candidates who completed successful immune tolerance induction (ITI) at least 5 years before screening are eligible, provided they have had no evidence of inhibitor recurrence (permanent or temporary) within 5 years prior to screening as may be indicated by detection of an inhibitor, FVIII half-life <6 hours, or FVIII recovery <66% since completing ITI.
* If human immunodeficiency virus (HIV)-positive at screening, have an adequate cluster of differentiation 4 (CD4) count (>200/mm3) and undetectable viral load (<50 genome copies [gc]/mL), are on an antiretroviral drug regimen, and have completed at least 12 weeks of this treatment regimen prior to screening.
* Meet the following inclusion criteria by cohort:

  * Cohort A: have documented history of prior treatment with FVIII prophylaxis (defined as receiving a prescribed dose and frequency of FVIII infusions with the intent to treat continuously for 52 weeks per year) for a minimum of 6 months prior to screening; and are willing to continue their FVIII prophylaxis during the Lead-In Period of this study (minimum of 24 weeks).
  * Cohort B: have documented history of prior treatment with FVIII on demand for a minimum of 6 months that shows ≥5 treated bleeds in the last 6 months prior to screening.
  * Cohort C: have documented history of prior treatment with emicizumab prophylaxis for a minimum of 6 months prior to screening.

Exclusion Criteria:

* Have an inherited or acquired bleeding disorder other than hemophilia A
* Have inherited or acquired thrombophilia, have signs of thromboembolic disease in the Investigator's judgment, or are on current treatment for thromboembolic disease. A history of previous catheter-associated thrombosis for which anti-thrombotic treatment is not currently ongoing is not considered an exclusion criterion.
* Have concurrent disease, treatment, or abnormality in clinical laboratory tests that could interfere with the conduct of the study or that would, in the opinion of the Investigator or Sponsor, preclude the candidate's safe participation in and completion of the study, or the interpretation of the study results.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-03-13 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2035-09-04 (Estimated)

PRIMARY OUTCOMES:
Annualized Bleed Rate (ABR) for All Bleeds [Cohort A] | Up to 66 weeks post-SPK-8011 infusion

SECONDARY OUTCOMES:
Median FVIII: C levels [Cohort A] | Up to approximately 10 years
ABR for treated bleeds [Cohort A] | Up to approximately 10 years
Percentage of Participants with ABR=0 for all bleeds; treated bleeds; treated spontaneous bleeds; and treated joint and target joint bleeds [Cohort A] | Up to approximately 10 years
ABR for treated spontaneous, joint, and target joint bleeds [Cohort A] | Up to approximately 10 years
Annualized FVIII dosage [Cohort A] | Up to approximately 10 years
Proportion of Resolved Target Joints [Cohort A] | Up to approximately 10 years
Mean Change of Total Hemophilia Joint Health Score [Cohort A] | Baseline, up to 66 weeks post-SPK-8011 infusion
FVIII:C levels over time [Cohort A] | Up to approximately 10 years
Mean ABR for all bleeds and treated bleeds [Cohort C] | Up to approximately 10 years
FVIII: C levels over time from Week 26 [Cohort C] | Up to approximately 10 years
Proportion of Participants Who Receive IV Methylprednisolone (IVMP) Prior to Week 8 (Early IVMP) [Cohorts A, B, C] | Up to approximately 10 years
Proportion of Participants Who Receive Secondary Oral Immunomodulation [Cohorts A, B, C] | Up to approximately 10 years
Median Time to First Immunomodulation-related Corticosteroid Dose [Cohorts A, B, C] | Up to approximately 10 years
Median Duration of Secondary Oral Immunomodulation [Cohorts A, B, C] | Up to approximately 10 years
Proportion of Participants with FVIII Inhibitor Development [Cohorts A, B, C] | Up to approximately 10 years
Proportion of participants with Treatment-related AEs of ALT Elevation [Cohorts A, B, C] | Up to approximately 10 years
Proportion of participants with treatment-related AEs of Infusion Reaction [Cohorts A, B, C] | Up to approximately 10 years
Number of participants with abnormal physical exam findings, abnormal vital signs, and abnormal selected clinical laboratory test results [Cohorts A, B, C] | Up to approximately 10 years
Proportion of participants with AEs and SAEs [Cohorts A, B, C] | Up to approximately 10 years
Proportion of participants with AESIs [Cohorts A, B, C] | Up to approximately 10 years

CONTACTS AND LOCATIONS:
Locations (27):
- United States (27):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Loma Linda University Health, Loma Linda, California
  - Orthopaedic Institute for Children/Orthopaedic Hemophilia Treatment Center, Los Angeles, California
  - Kaiser Permanente-Oakland Medical Center, Oakland, California
  - Kaiser Permanente-Roseville Medical Center, Roseville, California
  - Kaiser Permanente -Sacramento Medical Center, Sacramento, California
  - Kaiser Permanente -San Francisco Medical Center, San Francisco, California
  - University of California - San Francisco, San Francisco, California
  - Kaiser Permanente- Santa Clara Medical Center, Santa Clara, California
  - Kaiser Permanente-Vallejo Medical Center, Vallejo, California
  - Kaiser Permanente -Walnut Creek Medical Center, Walnut Creek, California
  - University of Florida, Gainesville, Florida
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Newark Beth Israel, Newark, New Jersey
  - Weill Cornell Medical Hospital, New York, New York
  - University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - University Hospitals Cleveland, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oregon Health & Sciences University, Portland, Oregon
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Cook Children's Hospital, Fort Worth, Texas
  - The University of Texas Health Science Center at Houston-Gulf States Hemophilia & Thrombosis Center, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Bloodworks NW, Seattle, Washington